CLINICAL TRIAL: NCT01591876
Title: The Effect of an Intra-dialytic Aerobic Exercise Intervention on Vascular Function in People Undergoing Maintenance Haemodialysis Therapy for Chronic Kidney Disease Stage 5. An Exploratory Study
Brief Title: Exercise and Vascular Function in Haemodialysis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: British Kidney Patients Association (Unknown)
Responsible Party: Principal Investigator, Sean Prescott, PhD Research Student, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/WS/0129
Record Dates: First submitted 2012-04-30; First posted 2012-05-04 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Kidney Disease Stage 5
Keywords: exercise; kidney disease; vascular function; haemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Kidney Diseases | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive muscle relaxation (Sham Comparator): As well as usual care participants in the control arm will receive instruction in progressive muscle relaxation.
  Interventions: Other: Progressive Muscle relaxation
- Aerobic exercise (Active Comparator): Intervention -moderate intensity aerobic exercise.
  Interventions: Other: Intradialytic aerobic exercise

INTERVENTIONS:
Other: Intradialytic aerobic exercise — Participants in the intervention group will undertake moderate intensity aerobic exercise. Exercise modality will be recumbent cycling during the first two hours of haemodialysis sessions. Exercise prescription is set using a graded exercise test and anchored to a perceived level of exertion using the BORG scale. Training stimulus is maintained by the participant by increasing the cycling resistance when perceived exertion drops by one point at the current resistance level. Adherence and training volume is recorded during the intervention period.
  Arms: Aerobic exercise
Other: Progressive Muscle relaxation — This is a sequence of stretching and relaxation of the major muscle groups of the body. Participants are initially given detailed information regarding the technique and then provided with a recorded version which they listen to for 30-40 minutes during dialysis sessions. Participants in this group are offered the exercise programme at the end of three months.
  Arms: Progressive muscle relaxation

SUMMARY:
The aim of this study is to evaluate whether a three month intra-dialytic exercise programme improves arterial function.

DETAILED DESCRIPTION:
Life expectancies in haemodialysis patients are significantly shorter than the general population due to higher cardiovascular disease risk. This is mediated by higher prevalence of cardiovascular risk factors associated with chronic kidney disease and the haemodialysis procedure. Consequently ageing of the arterial system is accelerated in this condition leading to higher prevalence of arterial plaques and increased arterial stiffness.

Higher physical activity and fitness are associated with lower cardiovascular disease and all-cause mortality in haemodialysis patients and the general population. Moreover, physical inactivity is associated with increased arterial stiffness and plaques which narrow heart arteries. Worryingly the haemodialysis population is on average highly inactive with low fitness.

Current research demonstrates that exercise which improves fitness improves arterial health. Increased bloodflow during exercise stimulates the release of nitric oxide causing arteries to dilate. Regular exercise is believed to lead to beneficial remodelling of arteries and lower arterial stiffness. Exercise is reported to improve arterial function across a range of conditions. However published research regarding the possible benefits of long term aerobic exercise on arterial health in this population is conflicting. Limitations in study design, moderately high participant dropout rates and low statistical power hamper a definitive conclusion. Importantly a gold standard measure of arterial function has not been used in previously published studies.

There is ample evidence that exercise programmes in people on dialysis improve fitness, physical function, and quality of life. It is also clear that a state of higher physical activity and fitness is associated with better arterial function in the general population. It would be advantageous for reasons of health counselling to determine whether the process of improving physical fitness and activity levels may also improve arterial health in haemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage 5 CKD patients (GFR <15 mL/min) receiving maintenance haemodialysis therapy
* Male or female
* Aged >18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Unstable cardiovascular conditions
* Recent cerebrovascular event
* Excess inter-dialytic weight gain
* Use of corticosteroids, anabolic therapies,
* Co-morbid catabolic conditions
* Serum potassium regularly >6mmol/L
* Recent pulmonary thromboembolism
* Psychiatric illness including anxiety, mood and untreated eating disorders
* Infection or course of antibiotics within one month of study period.
* Dementia or severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-07 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Brachial artery flow mediated dilatation | Baseline and 12 week follow-up
  Brachial artery diameter is measured using vascular ultrasound. A cuff similar to that used for blood pressure is then inflated around the forearm for 5 minutes. Following cuff release vascular ultrasound is used to measure arterial dilation in response to reactive hyperaemia. Relative change in diameter provides a measure of endothelial function. Images are recorded over a period of 4-5 minutes post cuff release.

SECONDARY OUTCOMES:
Aortic pulse wave velocity | Baseline and three month follow-up
  Aortic pulse wave velocity is measured using a Vicorder (Skidmore Medical, Bristol UK). Briefly the Vicorder measures the time taken for a pulse wave to travel between a pressure cuff located on the carotid artery and another at the site of the femoral artery. The calculated velocity of the pulse wave is a measure of central arterial stiffness.
Maximal aerobic power | Baseline and three months
  Peak aerobic power is assessed using a graded exercise test with respiratory gas analysis. An Astrand protocol will be used with cycle ergometry. Participants continue until volitional exhaustion or the test is terminated by the investigator. An oxygen uptake figure in ml/kg/min is a measure of peak aerobic power (VO2peak)
Timed up-and-go | Baseline and three month follow-up
  The time taken to stand up from a chair, walk three metres and return is recorded. This is a functional measure of mobility with a threshold time related to falls and fractures.
Sit-to-stand 5 | Baseline and 3 month follow-up
  The time taken to stand up from a chair five times without using upper limb assistance is recorded. This is a surrogate measure of lower limb power with a threshold that is related to balance and risk of falls.
Non exercise questionnaire | Baseline and 3 month follow-up
  A non-exercise questionnaire utilising anthropometry, gender and self reported physical activity will be used to estimate aerobic fitness. This method carries minimal burden compared to physical performance tests and is a useful screening tool for health counselling.
Physical activity | Baseline and 3 month follow-up
  Physical activity over a seven day period will be measured using an Actigraph accelerometer. The monitor measures body movement as activity counts which may be categorised according to level of intensity using established cut-points.
Kidney Disease Quality of Life Short Form (KDQOL) | Baseline and 3 month follow-up
  The KDQOL is a self-administered questionnaire designed to measure generic health related quality life as well as condition specific items. Higher scores indicate better quality of life.
Duke Activity Status Index | Baseline and 3 months
  This self administered 12 item questionnaire provides a self reported measure of physical capacity. Higher scores indicate higher fitness and ability to perform activities of daily living.
Leicester Uraemic Symptom Scale (LUSS) | Baseline and 3 month follow-up
  The LUSS provides a measure of condition related symptom burden. it records the number of symptoms, frequency and their level of intrusiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Mercer, Professor, Study Director — Queen Margaret University
Locations (1):
- Monklands Hospital, Airdrie, United Kingdom